CLINICAL TRIAL: NCT03433066
Title: Evaluation of Advanced Platelet-rich Fibrin in Management of Periodontal Intrabony Defects
Brief Title: Advanced Platelet Rich Fibrin in Periodontal Angular Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Jaylane kadry Ghonima, Instructor Jaylane Kadry Ghonima, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: platelet rich fibrin
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Intrabony Periodontal Defect
Keywords: advanced platelet-rich fibrin
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This clinical study will be conducted on twenty-two (22) interproximal intrabony defects in patients with moderate to severe chronic periodontitis.These patients will be divided randomly into two groups:
  * Group I: (test) will include eleven interproximal intrabony defects that will be treated with (Advanced platelet rich fibrin & biphasic alloplast)
  * Group II: (control) will include eleven interproximal intrabony defects that will be treated with (biphasic alloplast mixed with saline.)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Test) (Experimental): Advanced platelet-rich fibrin mixed with biphasic alloplast
  Interventions: Procedure: Advanced platelet-rich fibrin mixed with biphasic alloplast
- Group II (control) (Active Comparator): Biphasic alloplast mixed with saline
  Interventions: Procedure: Biphasic alloplast mixed with saline

INTERVENTIONS:
Procedure: Advanced platelet-rich fibrin mixed with biphasic alloplast — mucoperiosteal flaps will be reflected to expose the defects , which will be debrided properly and finally filled with the freshly prepared Advanced platelet-rich fibrin mixed with the biphasic alloplast.
  Arms: group I (Test)
Procedure: Biphasic alloplast mixed with saline — mucoperiosteal flap will be reflected to expose and clean the intrabony defect ,then it will be filled with biphasic alloplast mixed with saline.
  Arms: Group II (control)

SUMMARY:
The aim of this study is to clinically and radiographically evaluate the efficacy of advanced platelet-rich fibrin (A-PRF) when used with biphasic alloplast in the management of intrabony defects in patients with moderate to severe chronic periodontitis.

DETAILED DESCRIPTION:
Biphasic alloplasts have been successfully used in management of intrabony defects. Advanced platelet-rich fibrin is believed to contain higher amount of growth factors and white blood cells than the well known PRF. Although there are some studies on the use of PRF in the treatment of intrabony defects, to date none of them evaluate the effect of the A-PRF. Therefore, a randomized controlled clinical trial was conducted to compare the healing of intrabony defects treated with A-PRF/biphasic alloplast combination and to those obtained with biphasic alloplast mixed with saline. Using a parallel arm design, 22 intrabony defects were randomly treated with either biphasic alloplast mixed with saline (control group) or with A-PRF/ biphasic alloplast combination (test group). The following clinical parameters were recorded at baseline, three and six months postoperatively : plaque index (PI), modified gingival index (MGI), probing depth (PD), clinical attachment level (CAL), while these radiographic measurements were recorded at baseline and six months postoperatively: bone fill and bone density.

ELIGIBILITY:
Inclusion Criteria:

* They should be diagnosed as having moderate -severe chronic periodontitis according to the American Academy of Periodontology classification on gingival and periodontal diseases (1999)
* Clinical attachment loss (CAL) ,radiographic evidence of the presence of at least one intrabony defect.
* Patient's age between 25 to 55 years.
* Both sexes.
* No periodontal surgeries in the area of interest during the previous 6 months.
* The presence of intrabony defects (IBD) ≥3 mm deep (distance between alveolar crest and deepest point in the defect estimated from radiographs and confirmed upon surgical exposure).
* An interproximal probing depth (PD) ≥5 mm and clinical attachment loss (CAL) ≥3mm after phase I therapy in maxillary/ mandibular teeth.
* The presence of an adequate zone of keratinized gingiva at the facial aspect of the selected tooth.

Exclusion Criteria:

* Patients who could not maintain O'leary plaque index (54) ≤10% after phase I therapy.
* Aggressive periodontitis patients.
* Patients with systemic conditions known to affect the periodontal status, or, under medications known to affect the outcomes of periodontal therapy.
* Pregnancy/lactation.
* Smoking and tobacco use in any form.
* Non vital teeth and teeth with grade III mobility.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level change | Baseline , 3 and 6 months posoperatively
  The distance from cemento-enamel junction to the depth of the sulcus recorded by a periodontal probe at baseline , 3 and 6 months postoperatively

SECONDARY OUTCOMES:
Probing depth change: | Baseline , 3 and 6 months postoperatively
  The distance from the gingival margin to the depth of the sulcus recorded by a periodontal probe at baseline and 6 months postoperatively
Radiographic bone density | Baseline and 6 months postoperatively
  Measuring the bone density before and after the procedure using CBCT
Radiographic bone fill | Baseline and 6 months postoperatively
  The actual bone formation in the intrabony defect measured on a CBCT in comparison to the baseline CBCT

CONTACTS AND LOCATIONS:
Overall Officials: Mohy Eldin A. ElRashidy, Professor, Study Chair
Locations (1):
- Periodontology department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miron RJ, Fujioka-Kobayashi M, Bishara M, Zhang Y, Hernandez M, Choukroun J. Platelet-Rich Fibrin and Soft Tissue Wound Healing: A Systematic Review. Tissue Eng Part B Rev. 2017 Feb;23(1):83-99. doi: 10.1089/ten.TEB.2016.0233. Epub 2016 Oct 10. PMID 27672729
- [Background] Mazor Z, Horowitz RA, Del Corso M, Prasad HS, Rohrer MD, Dohan Ehrenfest DM. Sinus floor augmentation with simultaneous implant placement using Choukroun's platelet-rich fibrin as the sole grafting material: a radiologic and histologic study at 6 months. J Periodontol. 2009 Dec;80(12):2056-64. doi: 10.1902/jop.2009.090252. PMID 19961389
- [Background] Choukroun J, Diss A, Simonpieri A, Girard MO, Schoeffler C, Dohan SL, Dohan AJ, Mouhyi J, Dohan DM. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part V: histologic evaluations of PRF effects on bone allograft maturation in sinus lift. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):299-303. doi: 10.1016/j.tripleo.2005.07.012. PMID 16504861
- [Background] Perut F, Filardo G, Mariani E, Cenacchi A, Pratelli L, Devescovi V, Kon E, Marcacci M, Facchini A, Baldini N, Granchi D. Preparation method and growth factor content of platelet concentrate influence the osteogenic differentiation of bone marrow stromal cells. Cytotherapy. 2013 Jul;15(7):830-9. doi: 10.1016/j.jcyt.2013.01.220. PMID 23731763
- [Background] Dohan Ehrenfest DM, Del Corso M, Diss A, Mouhyi J, Charrier JB. Three-dimensional architecture and cell composition of a Choukroun's platelet-rich fibrin clot and membrane. J Periodontol. 2010 Apr;81(4):546-55. doi: 10.1902/jop.2009.090531. PMID 20373539
- [Background] Ajwani H, Shetty S, Gopalakrishnan D, Kathariya R, Kulloli A, Dolas RS, Pradeep AR. Comparative evaluation of platelet-rich fibrin biomaterial and open flap debridement in the treatment of two and three wall intrabony defects. J Int Oral Health. 2015 Apr;7(4):32-7. PMID 25954068
- [Background] Agarwal A, Gupta ND, Jain A. Platelet rich fibrin combined with decalcified freeze-dried bone allograft for the treatment of human intrabony periodontal defects: a randomized split mouth clinical trail. Acta Odontol Scand. 2016;74(1):36-43. doi: 10.3109/00016357.2015.1035672. Epub 2015 May 14. PMID 25972081